CLINICAL TRIAL: NCT02585271
Title: Transanal Decompression Tube Versus Stent as a Bridge to Surgery for Acute Malignant Left-sided Colonic and Rectal Obstruction
Brief Title: Transanal Decompression Tube Versus Stent for Acute Malignant Left-sided Colonic and Rectal Obstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We can not get enough sample size.
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46650455-0
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Colonic Cancer; Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transanal decompression tube (Other): Patients undergo placement of the transanal decompression tube as a bridge to surgery
  Interventions: Device: Transanal decompression tube
- Stent (Other): Patients undergo placement of the stent as a bridge to surgery
  Interventions: Device: Stent

INTERVENTIONS:
Device: Transanal decompression tube — 22 Fr transanal decompression tube
  Arms: Transanal decompression tube
Device: Stent — self-expandable colorectal nitinol alloys stent
  Arms: Stent

SUMMARY:
The purpose of this study is to compare the clinical outcomes of transanal decompression tube as a bridge to surgery with stent as a bridge to surgery for acute malignant left-sided colonic and rectal obstruction.

DETAILED DESCRIPTION:
Approximately 8-47 % of patients with colorectal cancer will present with colonic obstruction. Left-sided colonic and rectal cancer is responsible for nearly 70% of acute colonic obstruction. Emergency colonic surgery for acute obstruction is associated with a higher mortality and morbidity rate than elective surgery. Preoperative decompression results in a less dilated bowel that is more amenable to an elective surgery. Both transanal decompression tube and stent can serve a good preoperative decompression effect and serve a good bridge to surgery. Investigators aim to compare the clinical outcomes of transanal decompression tube as a bridge to surgery with stent as a bridge to surgery for acute malignant left-sided colonic and rectal obstruction.

ELIGIBILITY:
Inclusion Criteria:

1. definite diagnosis of left-side colonic or rectal obstruction;
2. symptomatic colonic obstruction for less than 1 week;
3. colonic obstruction caused by a histologically proven malignant colonic tumor

Exclusion Criteria:

1. suspected benign colonic or rectal obstruction;
2. right-side colonic obstruction;
3. patients with signs of peritonitis;
4. dysfunction of blood coagulation, active bleeding, active infection, and significant cardiac or pulmonary disease;
5. patients who do not want to undergo surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Creation of stoma | From the date of randomization until the date of first documented creation of stoma, assessed up to 24 months
  Creation of stoma include temporary and definitive stoma.

SECONDARY OUTCOMES:
Transanal decompression tube/stent-related complications | From the date of randomization until the date of first documented transanal decompression tube/stent-related complication, assessed up to 7 days
  Transanal decompression tube/stent-related complications usually include bowel perforation, migration, and stent re-obstruction.
Surgery-related complications | From the date of randomization until the date of first documented surgery-related complication, assessed up to 24 months
  Surgery-related complications usually include wound complications and anastomotic leak.
Overall survival | From the date of randomization until the date of death from any cause, assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tao Song, MD, Study Director — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu YS, Song T, Guo YT, Shao GQ, Du HT, Li DC, Fu YF. Placement of the Decompression Tube as a Bridge to Surgery for Acute Malignant Left-Sided Colonic Obstruction. J Gastrointest Surg. 2015 Dec;19(12):2243-8. doi: 10.1007/s11605-015-2936-7. Epub 2015 Sep 9. PMID 26354721